CLINICAL TRIAL: NCT02641431
Title: Electrical Substrate Elimination in Brugada Syndrome. Results in 135 Consecutive Patients
Brief Title: Epicardial Ablation in Brugada Syndrome
Acronym: BRUGADA_I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Carlo Pappone, MD, IRCCS Policlinico S. Donato
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR-01-2015
Record Dates: First submitted 2015-11-11; First posted 2015-12-29 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2017-11

CONDITIONS: Brugada Syndrome
Keywords: radiofrequency ablation; mapping; sudden death; syncope
MeSH Terms: conditions — Brugada Syndrome; Death, Sudden; Syncope | interventions — Ajmaline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- mapping/ablation (Experimental): Epicardial substrate identification consisted in mapping the entire RV epicardial surface under baseline conditions and after ajmaline infusion (1mg/kg in 5 minutes).We obtained 3 groups of RV epicardial maps using CARTO3 system: 1) bipolar/unipolar voltage map, 2) local activation time map (LAT), and 3) potential duration map (PDM), in which abnormal long-duration bipolar electrograms were defined as low-frequency (up to 100 Hz) prolonged duration (> 200 ms) bipolar signals with delayed activity extending beyond the end of the QRS complex. Epicardial ablation was performed during sinus rhythm using a stepwise strategy in a descending order of abnormal potential duration as displayed on the map and beginning from the longest potentials.
  Interventions: Procedure: mapping/ablation; Drug: Ajmaline; Procedure: ablation; Procedure: mapping

INTERVENTIONS:
Procedure: mapping/ablation — Mapping/ablation procedures will be performed under general anesthesia. After femoral venous access and percutaneous epicardial access, a multipolar catheter will be positioned at the right ventricle apex. High-density endocardial and epicardial electroanatomical maps will be performed using the CARTO3 system to define areas of delayed fragmented prolonged potentials during stable sinus rhythm and during spontaneous or ajmaline-induced type 1 BrS ECG pattern. Ajmaline (1mg/Kg in 5 minutes) will be used for the provocative test. Complete endo and epicardial maps will be obtained to ensure reconstruction of a 3-dimensional geometry of the cardiac chambers and to identify areas of abnormal electrograms as characterized by prolonged fragmented ventricular signals
  Other Names: voltage, activation and duration maps
Drug: Ajmaline — Epicardial mapping will be performed before and after ajmaline (1mg/Kg in 5 minutes).
  Other Names: Pharmacological testing
Procedure: ablation — Radiofrequency will be delivered on areas of the abnormal electrograms using an externally irrigated 3.5-mm tip ablation catheter.
  Other Names: RFA
Procedure: mapping — A re-map focusing on the targeted area will be obtained after ablation. Re-mapping and ajmaline reinfusion will be used to confirm the elimination of all the abnormal electrogram and BrS-ECG pattern disappearance.

SUMMARY:
This prospective study evaluates the methodology and results of epicardial mapping/ablation in a large series of consecutive selected BrS patients and to verify if RFA could normalize the consequences of a genetic disease.

DETAILED DESCRIPTION:
The present Registry is designed as a prospective, monocentric study. All patients referred to the Arrhythmology Department of IRCCS Policlinico San Donato Milanese, University- Hospital, for the management of BrS and fulfilling the selection criteria will be invited to participate in the study and will be asked their written consent to the participation in the trial.

Mapping and RFA procedure will be performed following a standardized procedure in hospital settings. Patients will be monitored for at least 3 days after procedure.

Before hospital discharge, echocardiography and 12-lead ECG will be performed in all patients. An ajmaline test will be systematically performed after the procedure and thereafter at 3, 6, and 12 months after ablation.

Patients will be followed up clinically after procedure as per normal clinical practice. Follow-up visits will be scheduled at 3, 6, and 12 months. 12-lead ECG and ICD interrogation will be performed at each follow-up visits. Patients will be instructed to immediately contact the center in case of symptoms suggestive of ventricular arrhythmias. Documentation for intercurrent events will be requested and collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by Brugada Syndrome, profiled by genetic testing, with documented spontaneous or drug-induced type I BrS ECG pattern, with symptoms attributable to ventricular arrhythmias and presenting multiple documented arrhythmic episodes
* Patients with an ICD already implanted
* Patients referred to the center for an electrophysiological study and indication to a potential concomitant radio-frequency catheter ablation (RFA) of ventricular arrhythmia or ventricular fibrillation
* Age ≥ 18
* Willingness to attend follow-up examinations
* Written informed consent to the participation in the trial

Exclusion Criteria:

* Pregnancy or breast-feeding
* Patients with low arrhythmic risk (Brugada pattern III)
* Life expectancy < 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Absence of the ECG Br pattern | 1 day
  Disappearance of the BrS-ECG pattern before and after ajmaline immediately after epicardial ablation and at discharge.

SECONDARY OUTCOMES:
Absence of episodes of ventricular arrhythmias | 3 months after procedure
  Absence of ECG Br pattern and arrhythmic episodes as documented by ICD interrogation, particularly in patients with worst clinical presentation and frequent ICD discharges
Absence of episodes of ventricular arrhythmias | 6 months after procedure
  Absence of ECG BR pattern and arrhythmic episodes as documented by ICD particularly in patients with worst clinical presentation and frequent ICD discharges.
Absence of episodes of ventricular arrhythmias | 12 months after procedure
  Absence of ECG Br pattern and arrhythmic episodes will be evaluated clinically as documented by ICD particularly in patients with worst clinical presentation and frequent ICD discharges.
Complications | 1 day
  Acute complications during and after the procedure will be evaluated clinically. Potential pericardial damage will be evaluated clinically and by Echocardiography.
Long-term complications | 3 months
  Long-term complications will be evaluated 3 months after the procedure clinically and by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pappone, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brugada P, Brugada J. Right bundle branch block, persistent ST segment elevation and sudden cardiac death: a distinct clinical and electrocardiographic syndrome. A multicenter report. J Am Coll Cardiol. 1992 Nov 15;20(6):1391-6. doi: 10.1016/0735-1097(92)90253-j. PMID 1309182
- [Result] Brugada J, Pappone C, Berruezo A, Vicedomini G, Manguso F, Ciconte G, Giannelli L, Santinelli V. Brugada Syndrome Phenotype Elimination by Epicardial Substrate Ablation. Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1373-81. doi: 10.1161/CIRCEP.115.003220. Epub 2015 Aug 19. PMID 26291334
- [Result] Nademanee K, Veerakul G, Chandanamattha P, Chaothawee L, Ariyachaipanich A, Jirasirirojanakorn K, Likittanasombat K, Bhuripanyo K, Ngarmukos T. Prevention of ventricular fibrillation episodes in Brugada syndrome by catheter ablation over the anterior right ventricular outflow tract epicardium. Circulation. 2011 Mar 29;123(12):1270-9. doi: 10.1161/CIRCULATIONAHA.110.972612. Epub 2011 Mar 14. PMID 21403098
- [Derived] Ciconte G, Santinelli V, Vicedomini G, Borrelli V, Monasky MM, Micaglio E, Giannelli L, Negro G, Giordano F, Mecarocci V, Mazza BC, Locati E, Anastasia L, Calovic Z, Pappone C. Non-invasive assessment of the arrhythmogenic substrate in Brugada syndrome using signal-averaged electrocardiogram: clinical implications from a prospective clinical trial. Europace. 2019 Dec 1;21(12):1900-1910. doi: 10.1093/europace/euz295. PMID 31647530
- [Derived] Pappone C, Ciconte G, Manguso F, Vicedomini G, Mecarocci V, Conti M, Giannelli L, Pozzi P, Borrelli V, Menicanti L, Calovic Z, Della Ratta G, Brugada J, Santinelli V. Assessing the Malignant Ventricular Arrhythmic Substrate in Patients With Brugada Syndrome. J Am Coll Cardiol. 2018 Apr 17;71(15):1631-1646. doi: 10.1016/j.jacc.2018.02.022. PMID 29650119
- [Derived] Pappone C, Brugada J, Vicedomini G, Ciconte G, Manguso F, Saviano M, Vitale R, Cuko A, Giannelli L, Calovic Z, Conti M, Pozzi P, Natalizia A, Crisa S, Borrelli V, Brugada R, Sarquella-Brugada G, Guazzi M, Frigiola A, Menicanti L, Santinelli V. Electrical Substrate Elimination in 135 Consecutive Patients With Brugada Syndrome. Circ Arrhythm Electrophysiol. 2017 May;10(5):e005053. doi: 10.1161/CIRCEP.117.005053. PMID 28500178